CLINICAL TRIAL: NCT00002208
Title: A Multicenter, Open-Label, Randomized, 24-Week Study to Compare the Safety and Activity of Indinavir Sulfate, 800 Mg q 8 h Versus 1,200 Mg q 12 h in Combination With Zidovudine and 3TC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 246M; 069-00
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-02

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; Indinavir; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Lamivudine; Stavudine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
To demonstrate that the antiviral activity and safety/tolerability of a test regimen of indinavir is equivalent to that of a control regimen of indinavir when each is coadministered with zidovudine (ZDV) (or stavudine, d4T) and lamivudine (3TC) for 24 weeks to protease inhibitor- and 3TC-naive HIV-1-seropositive patients. To characterize the steady-state pharmacokinetic profiles of indinavir, ZDV (or d4T), and 3TC in the presence of each other, for both the control and test regimen groups.

DETAILED DESCRIPTION:
Patients are randomized to 1 of 2 arms:

Arm A: Indinavir plus ZDV plus 3TC. Arm B: Indinavir (test dose) plus ZDV plus 3TC. NOTE: d4T may be substituted for zidovudine for toxicity management. Patients are stratified based on prior use of nucleoside analogs (naive vs experienced to ZDV, dideoxyinosine [ddI], dideoxycytidine [ddC], and d4T) and screening viral RNA results (lower than 50,000 copies/mL vs more than 50,000 copies/mL).

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 seropositive status.
* CD4 count greater than 100 cells/mm3.
* Viral RNA above 10,000 copies/mL.
* Consent from parent or guardian if less than 18 years of age.

Exclusion Criteria

Prior Medication:

Excluded:

* Prior therapy with protease inhibitors.
* Prior therapy with 3TC.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - LAC/USC Med Ctr, Los Angeles, California
  - Kaiser Med Ctr, San Francisco, California
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Washington Univ, St Louis, Missouri
  - Univ Hosp / SUNY at Stony Brook / AIDS TMT Unit, Stony Brook, New York
  - Allegheny Univ Hosp, Philadelphia, Pennsylvania
  - Pittsburgh Treatment Ctr / Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown Univ / Miriam Hosp, Providence, Rhode Island
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Washington / AIDS Clinical Trial Unit, Seattle, Washington

REFERENCES:
- [Background] Haas DW, Arathoon E, Thompson MA, de Jesus Pedro R, Gallant JE, Uip DE, Currier J, Noriega LM, Lewi DS, Uribe P, Benetucci L, Cahn P, Paar D, White AC Jr, Collier AC, Ramirez-Ronda CH, Harvey C, Chung MO, Mehrotra D, Chodakewitz J, Nguyen BY; Protocol 054/069 Study Teams. Comparative studies of two-times-daily versus three-times-daily indinavir in combination with zidovudine and lamivudine. AIDS. 2000 Sep 8;14(13):1973-8. doi: 10.1097/00002030-200009080-00013. PMID 10997402